CLINICAL TRIAL: NCT07291466
Title: Erhebung Von präoperativer Ängstlichkeit Und Bewertung Beruhigender Maßnahmen: Anonyme Patientenbefragung
Brief Title: Assessment of Preoperative Anxiety and Evaluation of Calming Interventions: Anonymous Patient Survey
Acronym: anti-anxiety
Status: Recruiting | Type: Observational
Sponsor: Vera Guttenthaler (Other)
Responsible Party: Sponsor-Investigator, Vera Guttenthaler, study coordinator, University of Bonn
Organization: University of Bonn (Other)
Other Study IDs: 2025-290-BO
Record Dates: First submitted 2025-11-20; First posted 2025-12-18 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Anxiety
Keywords: Operation; anxiety; pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to better understand the anxiety of patients before elective surgeries and to investigate which measures for calming are perceived as helpful or pleasant. Adult, German-speaking patients (≥18 years) in the elective surgical setting at UKB are invited to participate. It is planned that at least 400 patients will take part in the survey. The survey is conducted anonymously, voluntarily, and without the collection of personal data. This is a purely observational study without any intervention.

DETAILED DESCRIPTION:
Patients who come to the premedication outpatient clinic are invited in the waiting area to participate in this anonymous written survey. Participation is voluntary. The survey takes approximately 10-15 minutes. No personal data are collected.

Anxiety is assessed using the State-Trait Operation Anxiety (STOA) and the Amsterdam Preoperative Anxiety and Information Scale (APAIS) questionnaires.

To address anxiety reduction, various possible measures are listed, and patients are asked to check all the options they consider helpful and appropriate. They are also given the opportunity to add further suggestions that are not included in the list.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years),
* German-speaking patients
* elective surgical setting

Exclusion Criteria:

* emergency surgery
* Patients with documented psychiatric disorders or confusion
* Individuals admitted under a court or official mandate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult, German-speaking patients (≥18 years) in the elective surgical setting at UKB are invited to participate.
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Record patients' stated preferences related to anxiety management. | baseline
  using multiple-choice and open-ended responses

SECONDARY OUTCOMES:
Assess patients' preoperative anxiety | baseline
  Using the STOA questionnaire. The STOA evaluates anxiety on two levels: the long-term, personality-related tendency toward surgical anxiety (trait) and the current state of anxiety (state), with cognitive and affective components. The STOA-State scale includes 10 items rated on a 4-point scale from 0 ("Not at all") to 3 ("Very much"), yielding a total score of 0-30. The STOA-Trait scale includes 20 items rated from 0 ("Almost never") to 3 ("Almost always"), with a total score of 0-60.
Assess patients' preoperative anxiety | baseline
  Using APAIS questionnaire. The APAIS is a validated, brief instrument with 20 items, assessing anxiety related to anesthesia and the surgical procedure. Anxiety scores range from 4 (no anxiety) to 20 (high anxiety), and the total score ranges from 6 to 30.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bonn, Bonn, Germany